CLINICAL TRIAL: NCT01595568
Title: Prevention and Reduction of Alcohol and Drug Problems in a Clinical Psychiatric Youth Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Eveline Perrier-Ménard, MD, Master student, St. Justine's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CER CHU Ste-Justine 3435
Record Dates: First submitted 2012-05-03; First posted 2012-05-10 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Alcohol Abuse; Drug Abuse; Mood Disorder; Anxiety Disorder; Conduct Disorder
Keywords: Adolescents; Dual Diagnosis; Mental Disorders; Substance Use Problems; Prevention
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Mood Disorders; Anxiety Disorders; Conduct Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Learning to cope with your impulsivity (Experimental): Cognitive-behavioural intervention targeting impulsive personality
  Interventions: Behavioral: Personality-targeted interventions
- Learning to cope with your sensation seeking (Experimental): Cognitive behavioural intervention designed to help sensation seeking youth manage their need for stimulation and excitement.
  Interventions: Behavioral: Personality-targeted interventions
- Learning to cope with your anxiety sensitivity (Experimental): Cognitive behavioural intervention teaching anxiety sensitive youth to manager their sensitivity to threat and anxiety.
  Interventions: Behavioral: Personality-targeted interventions
- Learning to manage your negative thinking (Experimental): Cognitive behavioural intervention targeting pessimistic and negative thinking in hopeless youth
  Interventions: Behavioral: Personality-targeted interventions

INTERVENTIONS:
Behavioral: Personality-targeted interventions — Motivational and cognitive behavioural interventions targeting four personality profiles. 2 90 minute group sessions with personality-matched peers facilitated by a trained therapist and co-facilitator
  Other Names: Preventure; Adventure
  Arms: Learning to cope with your impulsivity
Behavioral: Personality-targeted interventions — Motivational and cognitive behavioural interventions targeting four personality profiles. 2 90 minute group sessions with personality-matched peers facilitated by a trained therapist and co-facilitator
  Other Names: Preventure; Adventure
  Arms: Learning to cope with your sensation seeking
Behavioral: Personality-targeted interventions — Motivational and cognitive behavioural interventions targeting four personality profiles. 2 90 minute group sessions with personality-matched peers facilitated by a trained therapist and co-facilitator
  Other Names: Preventure; Adventure
  Arms: Learning to cope with your anxiety sensitivity
Behavioral: Personality-targeted interventions — Motivational and cognitive behavioural interventions targeting four personality profiles. 2 90 minute group sessions with personality-matched peers facilitated by a trained therapist and co-facilitator
  Other Names: Preventure; Adventure
  Arms: Learning to manage your negative thinking

SUMMARY:
In adolescents, mental health problems are frequently associated with substance misuse, even considered a risk factor for alcohol abuse and dependence. This dual diagnosis tends to complicate the patient's treatment and prognosis by increasing, among others, substance use problems, reckless behaviours, relationships and school problems and suicidal thoughts. It is therefore critical to invest time and effort into developing an efficient approach to prevent and reduce substance use problems and offer these children a more global and optimal treatment.

A brief personality-targeted intervention was developed with students of Canadian and English high schools based on four personality factors known to be implicated in the vulnerability to adolescent alcohol misuse (Impulsivity, Anxiety Sensitivity, Negative Thinking and Sensation Seeking) (Conrod et al., 2006,2008, O'Leary-Barrett 2010).

By helping the adolescents to develop better adaptive behaviours, this cognitive-behavioural intervention proved to reduce binge drinking, quantity and frequency of use and substance use problems (Conrod et al., 2006,2011).

The purpose of this study is to assess the impact of this intervention if combined to a regular treatment in a youth psychiatric population.

60 patients aged 14-17 years of a Child and Adolescent psychiatric department will be screened for personality risk with self-report assessments including the Substance Use Risk Profile Scale. Participants will be randomly assigned to a personality matched cognitive-behavioural intervention or a no-intervention control.

The main outcome measures of this study are alcohol and illicit drug outcomes. Secondary measures include mental health symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Motive for psychiatric consultation
* Able to provide consent from parent/guardian for participation in the study

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Change in Binge drinking frequency | Baseline - 4months
Change in Drinking frequency | Baseline - 4 months
Change in Drinking quantity | Baseline - 4 months
Change in Drinking problems | Baseline - 4 months

SECONDARY OUTCOMES:
Change in Emotional and behavioural problems | Baseline - 4 months
  Psychiatric symptoms (depression, panic anxiety, antisocial behaviours), coping skills, motives for drinking, assessed using the Strengths and Difficulties Questionnaire, the Drinking Motives Questionnaire and the Brief Symptom Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada